CLINICAL TRIAL: NCT06075823
Title: Effectiveness and Safety of Edge-to-edge MItral vaLve Repair in Patients With Severe mitraL rEgurgitatioN aNd cardIac ATTR amyLoidosis
Brief Title: Edge-to-edge Mitral Valve Repair in ATTR-CM
Acronym: MILLENNIAL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Christian Nitsche, Principle Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1830/2023
Record Dates: First submitted 2023-09-27; First posted 2023-10-10 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Mitral Regurgitation; ATTR-Cardiomyopathy; Edge-to-Edge Mitral Valve Repair
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional (Experimental): TEER + Optimal Medical Therapy
  Interventions: Device: TEER; Other: Optimal Medical Therapy
- Control (Active Comparator): Optimal Medical Therapy alone
  Interventions: Other: Optimal Medical Therapy

INTERVENTIONS:
Device: TEER — transcatheter edge-to-edge mitral valve repair for significant mitral regurgitation
  Arms: Interventional
Other: Optimal Medical Therapy — optimal heart failure management of ATTR-CM

SUMMARY:
No previous study has evaluated the effectiveness of transcatheter edge-to-edge mitral valve repair (TEER) in patients with ATTR-associated cardiomyopathy (ATTR-CM) and significant mitral regurgitation, as this specific patient population was specifically excluded from previous large TEER trials. From a pathophysiological perspective, effective treatment of significant regurgitant volume and consecutive improvement of forward volume appears highly desirable in a condition with intrinsically low output. However, whether this translates into improved functional capacity, better quality of life, and better clinical outcomes compared to conservative heart failure management alone remains to be investigated.

DETAILED DESCRIPTION:
It is the aim of this trial to investigate the effectiveness of TEER therapy in patients with proven ATTR-CM and concomitant significant MR as compared to medical therapy alone. Effectiveness will be tested via hard clinical outcomes, biomarkers, functional capacity, and quality of life.

ELIGIBILITY:
Inclusion criteria (all must be present)

* Proven ATTR-CM
* Significant symptomatic MR (3+ or 4+ by independent echocardiographic core laboratory assessment)
* Subject has been adequately treated per applicable standards, including for coronary artery disease and heart failure (e.g., diuretics)
* New York Heart Association (NYHA) functional class II, III, or ambulatory IV
* Local heart team has determined that mitral valve surgery will not be offered as a treatment option, even if the subject is randomized to the control group
* Left ventricular ejection fraction ≥20%
* Anatomical feasibility for TEER as per discretion of the implanting investigator
* Age 18 years or older
* Subject or guardian agrees to all provisions of the protocol, including the possibility of randomization to the Control group and returning for all required post-procedure follow-up visits, and has provided written informed consent

Exclusion criteria (all must be absent)

* AL-associated cardiomyopathy
* Aortic or tricuspid valve disease requiring surgery or transcatheter intervention
* Severe right ventricular dysfunction
* Hemodynamic instability requiring inotropic support or mechanical heart assistance
* Leaflet anatomy which may preclude TEER, proper device positioning on the leaflets or sufficient reduction in mitral regurgitation by TEER
* Life expectancy <12 months due to non-cardiac conditions
* Prior mitral valve leaflet surgery or any currently implanted prosthetic mitral valve, or any prior transcatheter mitral valve procedure
* Echocardiographic evidence of intracardiac mass, thrombus or vegetation
* Active endocarditis or active rheumatic heart disease or leaflets degenerated from rheumatic disease (i.e., noncompliant, perforated)
* Active infections requiring current antibiotic therapy
* Transesophageal echocardiography (TEE) is contraindicated or high risk
* Pregnant or planning pregnancy within next 12 months
* Currently participating in another investigational device study that has not reached its primary endpoint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2027-12-12 (Estimated); Study Completion 2028-12-12 (Estimated)

PRIMARY OUTCOMES:
A hierarchical combination of all-cause mortality, cumulative frequency of cardiovascular-related hospitalization, change from baseline in NT-proBNP, and change from baseline in 6MWT through month 24 | 24 months
  Each subject will be compared to every other subject within a stratum over outcomes of all-cause mortality (death due to any cause), cumulative frequency of cardiovascular-related hospitalizations (number of times a subject is hospitalized for cardiovascular-related causes), change from baseline in NT-proBNP, and change from baseline in the total distance walked in 6 minutes (distance in meters).
  The hierarchical approach with the Finkelstein-Schoenfeld test will be applied and the test recognizes the greater importance of the mortality endpoint. Scores are transformed to -1, 0, +1. The alternative hypothesis is a subject in the TEER+OMT group will have a greater score than a subject in the placebo group.

SECONDARY OUTCOMES:
Evaluate effects of TEER on quality of life (QoL) through Month 24 | 24 months
  Change from Baseline to Month 24 as measured in the Kansas City Cardiomyopathy Questionnaire Overall Summary score (KCCQ-OS). The KCCQ is a 23-item questionnaire developed to measure health status and health-related quality of life in subjects with heart failure. Items include heart failure symptoms, impact on physical and social functions, and how their heart failure impacts their quality of life (QoL). An Overall Summary score can be derived from the physical function, symptom (frequency and severity), social function and quality of life domains. For each domain, scores are transformed to a range of 0-100 using the formula, 100*[(mean of questions actually answered) - 1]/4, in which higher scores reflect better health status. The Overall Summary score is the mean of the domains scores, range from 0 to 100, in which higher scores reflect better health status.
Technical, device, and procedural success of TEER (in the TEER group only) | 12 months
  Technical, device, and procedural success of TEER as defined according to the definitions of the Mitral Valve Academic Research Consortium (MVARC)

OTHER OUTCOMES:
Effects of TEER on echocardiographic markers | 24 months
  Changes in forward stroke volume, ejection fraction, global longitudinal strain, etc.
Effects of TEER on invasive haemodynamics (in the TEER group only) | 1 day
  Intraprocedural changes (pre- and post-TEER) in pulmonary pressures in the TEER-group

CONTACTS AND LOCATIONS:
Overall Officials: Christian Nitsche, MD, PhD, Principal Investigator — Medical University of Vienna

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stone GW, Lindenfeld J, Abraham WT, Kar S, Lim DS, Mishell JM, Whisenant B, Grayburn PA, Rinaldi M, Kapadia SR, Rajagopal V, Sarembock IJ, Brieke A, Marx SO, Cohen DJ, Weissman NJ, Mack MJ; COAPT Investigators. Transcatheter Mitral-Valve Repair in Patients with Heart Failure. N Engl J Med. 2018 Dec 13;379(24):2307-2318. doi: 10.1056/NEJMoa1806640. Epub 2018 Sep 23. PMID 30280640
- [Result] Dona C, Nitsche C, Koschutnik M, Heitzinger G, Mascherbauer K, Kammerlander AA, Dannenberg V, Halavina K, Rettl R, Duca F, Traub-Weidinger T, Puchinger J, Gunacker PC, Lamm G, Vock P, Lileg B, Philipp V, Staudenherz A, Calabretta R, Hacker M, Agis H, Bartko P, Hengstenberg C, Fontana M, Goliasch G, Mascherbauer J. Unveiling Cardiac Amyloidosis, its Characteristics, and Outcomes Among Patients With MR Undergoing Transcatheter Edge-to-Edge MV Repair. JACC Cardiovasc Interv. 2022 Sep 12;15(17):1748-1758. doi: 10.1016/j.jcin.2022.06.009. Epub 2022 Aug 22. PMID 36008266
- [Result] Chacko L, Karia N, Venneri L, Bandera F, Passo BD, Buonamici L, Lazari J, Ioannou A, Porcari A, Patel R, Razvi Y, Brown J, Knight D, Martinez-Naharro A, Whelan C, Quarta CC, Manisty C, Moon J, Rowczenio D, Gilbertson JA, Lachmann H, Wechelakar A, Petrie A, Moody WE, Steeds RP, Potena L, Riefolo M, Leone O, Rapezzi C, Hawkins PN, Gillmore JD, Fontana M. Progression of echocardiographic parameters and prognosis in transthyretin cardiac amyloidosis. Eur J Heart Fail. 2022 Sep;24(9):1700-1712. doi: 10.1002/ejhf.2606. Epub 2022 Jul 27. PMID 35779241
- [Result] Nitsche C. Echocardiographic tracking of transthyretin cardiomyopathy: which parameters matter the most? Eur J Heart Fail. 2022 Sep;24(9):1713-1715. doi: 10.1002/ejhf.2639. Epub 2022 Aug 12. No abstract available. PMID 35906799